CLINICAL TRIAL: NCT07037927
Title: Minnesota Retaining Employment and Talent After Injury/Illness Network (RETAIN) Phase 3
Brief Title: Minnesota RETAIN Phase 3
Acronym: MN RETAIN
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mayo Clinic (Other)
Collaborators: Minnesota Department of Employment and Economic Development (Unknown); U.S. Department of Education (U.S. Federal Agency)
Responsible Party: Principal Investigator, Laura E. Breeher, Principal Investigator, Mayo Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 24-013097; H421F240147 (Other Grant/Funding Number: Department of Education)
Record Dates: First submitted 2025-06-17; First posted 2025-06-26 (Actual); Last update posted 2025-10-30 (Actual); Status verified 2025-10

CONDITIONS: Injuries Related Work; Illness Related Work; Disability
Keywords: RETAIN; Minnesota RETAIN; MN RETAIN; Illness Recovery; Injury Recovery; Out of work help; Work Placement assistance; Job Help; Work Help; Help Keeping my job; Stay at work; Return to work

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Phase 3 (Experimental): Individuals will be assigned a dedicated Minnesota RETAIN Return-to-Work Case Manager. Participants will be referred for additional career and workforce development resources when needed.
  Interventions: Other: RETAIN Program

INTERVENTIONS:
Other: RETAIN Program — Facilitates early intervention strategies to support workers in staying-at or returning-to-work (SAW/RTW) after injury or illness and preventing unnecessary disability. This is done by incorporating a Return-to-Work Case Manager as a member of the healthcare clinical team who acts as a liaison for the patient and assists in coordination of referrals between healthcare and Workforce Development services. Return-to-Work Case Managers will interact with treating providers of Minnesota RETAIN participants to ensure functionally based work restrictions are documented and shared with the patient's employer.

SUMMARY:
MN RETAIN Phase 3 is a non-randomized trial to evaluate the impact of RETAIN program expansion and services on workforce retention and reduction of future workplace disability in the state of MN. The program is funded by US Department of Education (DOE). There will be collaboration between partners to implement best practices in early intervention to support injured or ill employees in stay-at-work and return-to-work. MN RETAIN involves a partnership between Mayo Clinic and MN Department of Employment and Economic Development (DEED), and stakeholders throughout MN. MN DEED serves as the main recipient and administrator of the funding within the state with Mayo Clinic a subrecipients of the grant.

ELIGIBILITY:
Inclusion Criteria:

* > 18-years-old,
* MN Resident,
* Works or intends to work in MN,

Meets one of the following:

* Employed at the time of enrollment (must be a W2 employee) OR,
* Unemployed and in the workforce (looking for a job) referred by either:
* Dislocated Worker (DW) Program,
* Healthcare provider/care team managing work restrictions
* Within 6 months of last day of work,

Meets one of the following:

* Provider work restrictions of unable to work for at least 2 weeks
* Per healthcare team anticipated to be unable to work for at least 2 weeks
* Employer's inability to accommodate current work restrictions

Meets one of the following:

* Diagnosis of a personal injury or illness that impacts employment (acute injury/illness or exacerbation of a chronic condition).
* Surgery or procedure anticipated within the next 4-weeks that impacts employment
* Documentation of work restrictions (i.e., written note/form documentation in electronic medical record prior to enrollment)

Exclusion Criteria:

* Does not have the capacity to give appropriate informed consent,
* Active workers' compensation claim relating to the qualifying injury or illness,
* Pending application OR Receiving Social Security Disability Insurance (SSDI) or -Supplemental Security Income (SSI),
* Self-Employed (i.e., 1099 worker)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-07-07 (Actual); Primary Completion 2028-03-31 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Workers to maintain employment | 6 month after enrollment
  Of the individuals participating, the number who achieve or maintain competitive integrated employment at the end of the enrollment period.

SECONDARY OUTCOMES:
Engagement Statewide | 3 years
  Percentage of participants living in individual MN counties with a goal of at least 50% of counties.

OTHER OUTCOMES:
Accessibility for individuals with disabilities acutely impacting work based | 4 years
  Total number of categories of disabilities based on workforce innovation act categories

CONTACTS AND LOCATIONS:
Overall Officials: Laura Breeher, M.D, M.P.H, Principal Investigator — Mayo Clinic; Clayton Cowl, M.D, MS, Principal Investigator — Mayo Clinic
Locations (1):
- Mayo Clinic Rochester, Rochester, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No